CLINICAL TRIAL: NCT02269501
Title: The Effect of a Specific Exercise Program on Patients Suffering From Migraine and Co-existing Tension-type Headache and Neck Pain
Brief Title: Exercise in Migraine and Co-existing Tension-type Headache and Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Lotte Skytte Krøll, PT, MPH, PhD student, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2011-090
Record Dates: First submitted 2014-07-10; First posted 2014-10-21 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Migraine; Tension-type Headache; Neck Pain
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise treatment (Experimental): Exercise treatment
  Interventions: Other: Exercise treatment
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Other: Exercise treatment
  Arms: Exercise treatment

SUMMARY:
The purpose of this study is to study the effect of a physical exercise program on patients suffering from migraine and co-existing tension-type headache and neck pain. The investigators hypothesized that migraine patients are ofte physically inactive because of their headache and that they will benefit from a specific exercise program.

DETAILED DESCRIPTION:
Migraine and tension-type headache are among the most common neurological diseases and are causing reduced quality of life, private and socio-economic consequences in terms of medical consumption and work-related absenteeism. The clinical experience shows that physical activity, like cycling and brisk walking, can prevent migraine attacks, but the evidence of the efficacy is sparse.

The primary aim of the study is to investigate the acute and the long term effect of exercise on patients suffering from migraine and co-existing tension-type headache and neck pain.

The project will be the first of its kind that explores the effect of an exercise program on patients who both suffer from migraine, tension-type headache and neck pain. We expect that the participants from the exercise program will achieve a reduced pain impact on everyday life, an improved fitness and quality of life, and a decrease of absence days and medication use.

ELIGIBILITY:
Inclusion Criteria:

* Migraine
* Tension-type headache
* Neck pain

Exclusion Criteria:

* Whiplash injury or other significant neck trauma
* Nerve root compression
* Post traumatic headache
* Medication overuse headache
* Cluster headache
* Trigeminal neuralgia
* Pregnancy and breast feeding
* Severe physical and psychological illnesses
* Alcohol and or drug abuse
* Current insurance claim owing to headache
* Persons not able to speak or understand Danish
* Persons deemed not to implement the program because of musculoskeletal pain or physical limitations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-11; Primary Completion 2016-09 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Changes in pain | At baseline and after three, six and 12 months follow-up
  Pain intensity, pain frequency and pain duration for migraine, tension-type headache and neck pain based on four-weeks headache and neck pain diaries prior inclusion; and diaries filled out each day for three months during intervention and again four weeks prior to six months follow-up and again four weeks prior to 12 months follow-up

SECONDARY OUTCOMES:
Changes in headache and neck pain impact | At baseline and after three, six and 12 months follow-up
  Headache and neck pain impact measured by the following questionnaires: Impact of Migraine, Tension-Type Headache and Neck Pain (a newly developed questionnaire), International Physical Activity Questionnaire (IPAQ short form), Migraine Specific Quality of Life Questionnaire (MSQ v. 2.1), Psychological well-being index (WHO-5), Major Depression Inventory (MDI) and Neck Disability Index (NDI).
Changes in quatitative sensory testing | At baseline and after three and six months follow-up
  Quantitative sensory tests are measured by: Total tenderness score, local tenderness score, pressure pain threshold and suprathreshold pain sensitivity
Changes in aerobic fitness | At baseline and after three and six months follow-up
  Åstrands submaximal bicycle test

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Department of Neurology, Glostrup Municipality, Denmark